CLINICAL TRIAL: NCT01538277
Title: A Pilot Study of a Contact Force Catheter for Pulmonary Vein Antrum Isolation (CFC-PVAI)
Brief Title: A Pilot Study of a Contact Force Catheter for Pulmonary Vein Antrum Isolation
Acronym: CFC-PVAI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CFC-PVAI
Record Dates: First submitted 2012-02-20; First posted 2012-02-24 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2012-03

CONDITIONS: Atrial Fibrillation; Burden of Atrial Fibrillation
Keywords: contact force catheter; loop recorder
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Contact Force arm (Experimental): the real-time contact force will be known to the operator
  Interventions: Procedure: Contact Force during ablation
- Standard (Active Comparator): Standard ablation arm
  Interventions: Other: Standard ablation procedure

INTERVENTIONS:
Procedure: Contact Force during ablation — Radio Frequency Ablation procedure with real-time contact force information known to the operator
  Arms: Contact Force arm
Other: Standard ablation procedure — Standard ablation procedure
  Arms: Standard

SUMMARY:
The knowledge of the real-time contact force leads to a greater reduction in atrial fibrillation burden after pulmonary vein antrum isolation.

DETAILED DESCRIPTION:
A randomized controlled study comparing pulmonary vein antrum isolation with and without the knowledge of the real-time contact force. In both groups, a catheter, which is able to measure contact force (SmartTouch, ThermoCool catheter, Biosense Webster) will be used. In the control group, the operator will be blinded to the measured contact-force. In all patients, the ablation will be guided by a circumferential mapping catheter (Lasso, Biosense Webster), CARTO 3 mapping system and ablation of adenosine-induced reconnection will be performed in all patients. Follow-up will be performed by continuous monitoring using an implantable loop recorder (Reveal XT, Medtronic Inc, Minneapolis, Minn)

ELIGIBILITY:
Inclusion Criteria:

* Patients <75 years of age with atrial fibrillation who have had at least two episodes of symptomatic paroxysmal or short-lasting persistent atrial fibrillation in the foregoing 12 months undergoing the first pulmonary vein antrum isolation can be included.
* Patients having also persistent episodes of atrial fibrillation of shorter duration (the longest atrial fibrillation episode 3 months) on top of paroxysmal episodes will be included

Exclusion Criteria:

* Contraindication to anticoagulation treatment with vitamin K antagonists Amiodarone therapy Expected surgery for structural heart disease within the follow-up period Significant mitral valve disease NYHA III-IV Left ventricular ejection fraction < 35% Left atrial diameter > 5 cm Secondary atrial fibrillation (e.g. post-surgery, infections, hyperthyroidism) Age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-02; Primary Completion 2014-09 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Reduction in atrial fibrillation burden (after 3 months blanking period) in comparison with the period prior to ablation in the absence of antiarrhythmic drugs | 12 month follow after the RFA treatment
  The atrial fibrillation burden defined as the percentage of time spent i atrial fibrillation monitored by an implantable cardiac loop recorder.

SECONDARY OUTCOMES:
Contact Force distribution during procedure (g/cm2) Post ablation A-fib burden(% of time in atrial fibrillation) Complications (number) Time spent on RFA of each pulmonary vein (min.) Reconnected pulmonary veins during adenosine/isoprenaline | 12 month follow up after the RFA treatment

CONTACTS AND LOCATIONS:
Overall Officials: Henrik k Jensen, phD, Dr Med, Study Director — University of Aarhus
Locations (1):
- Aarhus University Hospital - Skejby, Aarhus, Denmark, Denmark